CLINICAL TRIAL: NCT04795895
Title: Ultrasound for Confirmation of Gastric Tube Placement in Critically Ill Patients Under Invasive Mechanical Ventilation, a Randomization Trial
Brief Title: Ultrasound for Confirmation of Gastric Tube Placement in Critically Ill Patients Under Invasive Mechanical Ventilation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No obvious difference of primary outcome was detected when external reviewing
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 201907167RINB
Record Dates: First submitted 2021-03-10; First posted 2021-03-12 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Ultrasound for Confirmation of Gastric Tube Placement in Critically Ill Patients Under Invasive Mechanical Ventilation
Keywords: Point-of-care ultrasound,ultrasound
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasonography (US) (Experimental)
  Interventions: Diagnostic Test: ultrasonography (US)
- Standard routine (SR) (Active Comparator)
  Interventions: Diagnostic Test: Standard routine (SR)

INTERVENTIONS:
Diagnostic Test: ultrasonography (US) — US evaluation was performed after insertion of the tube via subxiphoid approach for tube passing esophagogastric (EG) junction. The tube insertion procedure will be repeated no more than three attempts if no visualization by US.
  Arms: ultrasonography (US)
Diagnostic Test: Standard routine (SR) — Standard routine (SR)
  Arms: Standard routine (SR)

SUMMARY:
Introduction: Data using ultrasonography to confirm correct position of the gastric tube is heterogeneous in approach sites, combination exams, and methodology.

Aim: Find the best strategy to confirm gastric tube placement to avoid immediate complication.

Method: A randomized controlled trial was initiated to compare ultrasonography and standard routine method, using non-inferiority design. The study will be conducted in one medical ICU with 59 beds at a medical center. The primary outcome is the correct rate as comparing with the chest radiography in each group. Total 190 patients is needed with estimated 10% drop-out rate.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication of nasogastric tube placement
* Age than 20 years old.

Exclusion criteria:

* Facial trauma or head-base fractures
* Esophageal or gastric resection
* Esophageal strictures or alkaline injury
* Open wound in the area to prevent ultrasonography

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
correct rate as comparing with the chest radiography in each group | 1 day

SECONDARY OUTCOMES:
procedure time, tube placement confirmation time other than chest radiography method, and additional auscultation method in US group | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Chun Chien, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Test2, Taiwan